CLINICAL TRIAL: NCT01527331
Title: A ProspectiveTrial Using Video Images in Advance Care Planning in Hospitalized Seriously Ill Patients With Advanced Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011P000010
Record Dates: First submitted 2012-01-26; First posted 2012-02-07 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): usual care
- Video decision aid arm (Experimental)
  Interventions: Behavioral: video decision aid

INTERVENTIONS:
Behavioral: video decision aid — cpr video decision aid
  Arms: Video decision aid arm

SUMMARY:
The purpose of this study is to compare the decision making of hospitalized subjects with advanced cancer having a verbal discussion about CPR compared to subjects using a video.

DETAILED DESCRIPTION:
Aim 1: To recruit 150 subjects with advanced cancer admitted to the inpatient oncology ward with an overall prognosis of one year or less and randomly assign these subjects to:

1. a video visually depicting CPR preferences or
2. the current standard of care without the use of video (control).

Hypothesis 1: It is feasible to recruit and randomize 150 hospitalized subjects with advanced cancer and an overall prognosis of one year or less.

Aim 2: To compare the care preferences for CPR and intubation among subjects randomized to video and subjects randomized to the current standard of care without the video.

Hypothesis 2: Subjects randomized to the video intervention will be significantly more likely to opt against CPR and intubation compared to those who do not see the video.

Aim 3: To compare code-status documentation in the electronic medical records between subjects randomized to the video and those who are receiving the current standard of care without the video.

Hypothesis 3: Subjects randomized to the video are more likely to have their code status documented in the electronic medical records compared to those who do not see the video.

Aim 4: To compare the decisional conflict of subjects randomized to video and subjects randomized to the current standard of care without the video.

Hypothesis 4: When compared to subjects randomized to the current standard of care, subjects in the video intervention group will have lower decisional conflict (lower decisional conflict scores) when asked to choose CPR and intubation preferences.

Aim 5: To compare knowledge assessment of CPR of subjects randomized to video and subjects randomized to current standard of care without the video.

Hypothesis 5: When compared to subjects randomized to the current standard of care, subjects in the video intervention group will have higher knowledge assessment scores when asked questions regarding their understanding of CPR.

Aim 6: To compare code-status (CPR, and intubation) preferences in the electronic medical record on future hospitalizations up to one year post-hospital discharge of subjects randomized to video and subjects randomized to current standard of care without the video.

Hypothesis 6: Subjects randomized to the video are more likely to opt against CPR and intubation in the future compared to those who do not see the video.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects will be identified by the research assistant. The specific eligibility criteria include:

  1. Over the age of 60
  2. The ability to provide informed consent
  3. The ability to communicate in English
  4. An established diagnosis of metastatic cancer with a prognosis of one year or less confirmed with the attending physician on service.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
preferences for medical care regarding CPR (yes, no or unsure) | within 5 minutes of surveyor asking the questions

SECONDARY OUTCOMES:
knowledge of CPR | 5 minutes after the surveyor asks questions
  Knowledge of CPR will be ascertained using True/False questions and one multiple choice question. Answers will be tallied into a score. Subjects will answer questions before the intervention (Baseline) as well as immediately after the intervention (within approximately 15 minutes of the intervention).
code status on subsequent admissions (Full code, DNR/DNI, etc.) | subsequent hospital admissions within one year

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States